CLINICAL TRIAL: NCT06924463
Title: Identification de Signatures moléculaires spécifiques Dans le Rhabdomyosarcome de l'Enfant, de l'Adolescent et du Jeune Adulte, Par Analyse Spatiale du protéome Par spectrométrie de Masse
Brief Title: Identification of Specific Molecular Signatures in Pediatric, Adolescent, and Young Adult Rhabdomyosarcoma Through Spatial Proteome Analysis Using Mass Spectrometry
Acronym: AERO-RMS
Status: Recruiting | Type: Observational
Sponsor: Lille University (Other)
Collaborators: Centre Oscar Lambret, Lille, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: D2024-7
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Rhabdomyosarcoma
Keywords: rhabdomyosarcoma; molecular signatures; spatial proteome; targeted therapy
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: None AHT — This study does not involve any interventions. It analyzes pre-existing biological samples (FFPE tumor tissue) and clinical data from patients with rhabdomyosarcoma.

SUMMARY:
This non-interventional study aims to develop spatial proteomics for analyzing small FFPE tumor samples in rhabdomyosarcoma. It will identify molecular signatures linked to tumor regions, subtypes, survival, and treatment resistance, using pre-existing samples and data.

DETAILED DESCRIPTION:
This is a non-interventional, monocentric, retrospective cohort study aimed at developing a spatial proteomics analysis method for small tumor samples (FFPE) to precisely characterize proteins at the tissue level in rhabdomyosarcoma (RMS). Using mass spectrometry, the study will identify molecular signatures associated with different tumor regions, histological subtypes, patient survival, and treatment resistance. The goal is to identify potential protein biomarkers and therapeutic targets. Data from clinical samples will be analyzed to find biomarkers correlated with survival and resistance to treatment. No patient intervention is required, as the study uses pre-existing biological samples and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 25 years at the time of initial diagnosis
* Diagnosis of rhabdomyosarcoma confirmed histologically
* Care at the Oscar Lambret Center between January 2005 and November 2024
* No objection to the re-use of data and biological samples collected as part of care for research activities.

Exclusion Criteria:

* Unavailability of biological sample in FFPE from biopsy and/or surgical specimen for diagnosis at Centre Oscar Lambret;
* Patient under guardianship or trusteeship.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Oscar Lambret Center (Lille, France)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Spatial Proteomic Profiling of Tumor Samples | 12 months (study duration)
  Evaluate the ability to obtain distinct proteomic profiles from at least 75% of tumor samples analyzed, with a minimum of two distinct profiles identified per sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Oscar Lambret Center, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No